CLINICAL TRIAL: NCT07398547
Title: The Effect of Training Frequency on Explosive Strength in Adolescent Tennis Players During a Six-Week Functional Training Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, alyildirim, PhD, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1071
Record Dates: First submitted 2026-01-24; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Exercise Therapy
Keywords: adolescent tennis players; explosive strength; performance development; functional training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Our study is designed as a prospective, two-group experimental study. Participants will be randomly assigned to two groups: the first group will participate in a 60-minute functional training program once a week, and the second group will participate in a 60-minute functional training program three times a week. At the end of the six-week program, the effects of training frequency will be assessed by comparing changes in explosive strength performance across groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Frequency Functional Training Group (LFFT) (Other): Participants in this group performed the functional training program once per week for six consecutive weeks. Each session lasted approximately 60 minutes and included dynamic warm-up, multi-joint functional exercises, and cool-down activities supervised by the same physiotherapist.
  Interventions: Other: Low-Frequency Functional Training Group (LFFT)
- High-Frequency Functional Training Group (HFFT) (Experimental): Participants in this group performed the same functional training program three times per week for six consecutive weeks. Each 60-minute session followed the same structure as the low-frequency program and was conducted under identical supervision and environmental conditions.
  Interventions: Other: High-Frequency Functional Training Group (HFFT)

INTERVENTIONS:
Other: High-Frequency Functional Training Group (HFFT) — Participants in this group performed the same functional training program three times per week for six consecutive weeks. Each 60-minute session followed the same structure as the low-frequency program and was conducted under identical supervision and environmental conditions.
  Other Names: exercise
  Arms: High-Frequency Functional Training Group (HFFT)
Other: Low-Frequency Functional Training Group (LFFT) — Participants in this group performed the same functional training program once per week for six consecutive weeks. Each 60-minute session followed the same structure as the low-frequency program and was conducted under identical supervision and environmental conditions.
  Other Names: exercise
  Arms: Low-Frequency Functional Training Group (LFFT)

SUMMARY:
Adolescence is a period characterized by rapid growth and development, characterized by intense structural, functional, and neuromuscular changes in the musculoskeletal system. The rapid height growth and proportional changes that occur during this period can negatively impact athletic performance by disrupting muscle strength and flexibility. Deficiencies in lower extremity muscle strength, in particular, can lead to decreased performance and increased injury risk in sports requiring high agility, balance, and explosive power, such as tennis.

Functional training programs are holistic exercise approaches that aim to improve neuromuscular control, balance, coordination, and muscle strength by simultaneously training multiple muscle groups. This type of training is particularly important in adolescent athletes because it supports the development of strength, endurance, and explosive power. Training frequency, in turn, plays a decisive role in muscle adaptation and performance enhancement by influencing the balance between loading and recovery.

Literature contains limited studies directly examining the effects of functional training frequency on explosive power performance in young athletes. Most existing research has focused on adult or professional athletes, and experimental studies comparing the effects of different training frequencies in adolescent tennis players are insufficient.

In this context, the aim of our study was to examine the effects of a six-week functional training program implemented at different training frequencies on lower extremity explosive strength parameters in adolescent tennis athletes.

DETAILED DESCRIPTION:
Adolescence is a dynamic period accompanied by rapid growth and development, characterized by intense structural, functional, and neuromuscular changes in the musculoskeletal system. During this period, weakness in the lower extremity muscles can lead to decreased performance and increased injury risk in sports requiring agility, balance, and explosive power, such as tennis.

Functional training programs are comprehensive exercise approaches that improve neuromuscular coordination, balance, and stabilization by simultaneously activating multiple muscle groups. These types of training are particularly important for young athletes because they support sport-specific movement patterns, increase muscle strength, and optimize the energy transfer chain. Training frequency is a key variable in determining muscle adaptation, recovery time, and load balance. Therefore, studies examining the effects of different training frequencies on explosive power development in young tennis athletes are of great scientific and practical value.

Healthy adolescent tennis players who volunteer to participate will be included in the study. After recording demographic and sport-specific information, participants' explosive strength performance will be assessed using the Countermovement Jump (CMJ), Squat Jump (SJ), Single Leg Jump (SLJ), and Reactive Strength Index (RSI) tests. Participants will be randomly assigned to two groups: the first group will participate in a 60-minute functional training program once a week, and the second group will participate in a 60-minute functional training program three times a week. The programs will last six weeks, and all sessions will be conducted by the same physiotherapist. Assessments will be conducted before and after the six-week training program. The study employed a two-group, pretest-posttest design. This study aims to demonstrate the effects of different training frequencies on explosive strength development in adolescent tennis athletes, contributing to the scientific basis of training plans for young athletes and to optimize performance.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent tennis players aged 12-18 years.
* Have at least two years of regular tennis training history.
* Regularly practice tennis at least three days a week.
* Have not had an acute injury or surgery affecting the lower extremities in the last six months.
* Have the physical ability to fully complete explosive strength tests (CMJ, SJ, SLJ, RSI).
* Individuals who voluntarily agreed to participate in the study and provided written consent from their parents.

Exclusion Criteria:

* Those with ongoing pain, instability, or deformity in the knee, hip, ankle, or spine area.
* Those who have undergone a musculoskeletal physical therapy or rehabilitation program within the last 6 months.
* Those with a systemic disease that may affect neurological, vestibular, or balance.
* Those who experience pain or fatigue to the extent that they cannot complete postural analysis or performance tests.
* Those who do not have a regular sports history or have not trained regularly in the last 3 months.
* Participants who exhibited a lack of cooperation during the assessment process that could compromise measurement consistency.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Countermovement Jump Test (CMJ) | 6 weeks
  The participant performs a rapid squat from an upright position with hands on hips, followed by a maximum vertical jump. This assesses lower extremity explosive strength and elastic energy utilization.
Squat Jump (SJ) Test | 6 weeks
  The participant is fixed in a position of approximately 90° flexion of the knee and hip joints, then performs a maximum vertical jump without using the arms. It measures pure concentric muscle strength.
Reactive Strength Index (RSI) Test | 6 weeks
  It's typically performed using a drop jump protocol. The participant jumps onto the platform from a specific height and bounces back up as quickly as possible after contact with the ground. RSI is calculated based on jump height and ground contact time; it measures reactive strength and stretch-shortening cycle (SSC) effectiveness.
Standing Long Jump (SLJ) Test | 6 weeks
  The participant stands with their feet parallel and jumps as far forward as possible using their arms. Lower extremity explosive strength is assessed by measuring the jump distance.
Assessment of normal joint motion | 6 weeks
  The Normal Joint Motion Assessment (NJM) Test is an objective method used to measure joint range of motion. In the study, participants' hip and knee joint flexion and extension angles will be assessed using the NJM test using a universal goniometer. Measurements will be made using active range of motion, and each measurement will be repeated three times and averaged.

CONTACTS AND LOCATIONS:
Locations (1):
- Sportplus Tennis Academy, Istanbul, Maltepe, Turkey (Türkiye)

REFERENCES:
- [Result] Axman S, Stausholm MB, Volk NR, Ferrauti A, Magnusson SP, Couppe C. Physical Performance Tests in 8008 Competitive Youth Tennis Players-A Systematic Review and Meta-Analysis of Normative Values. Eur J Sport Sci. 2025 Sep;25(9):e70023. doi: 10.1002/ejsc.70023. PMID 40884448
- [Result] Colomar J, Baiget E, Corbi F. Influence of Strength, Power, and Muscular Stiffness on Stroke Velocity in Junior Tennis Players. Front Physiol. 2020 Mar 6;11:196. doi: 10.3389/fphys.2020.00196. eCollection 2020. PMID 32210838
- [Result] Myer GD, Faigenbaum AD, Ford KR, Best TM, Bergeron MF, Hewett TE. When to initiate integrative neuromuscular training to reduce sports-related injuries and enhance health in youth? Curr Sports Med Rep. 2011 May-Jun;10(3):155-66. doi: 10.1249/JSR.0b013e31821b1442. PMID 21623307
- [Result] Fernandez-Fernandez J, Ulbricht A, Ferrauti A. Fitness testing of tennis players: how valuable is it? Br J Sports Med. 2014 Apr;48 Suppl 1(Suppl 1):i22-31. doi: 10.1136/bjsports-2013-093152. PMID 24668375
- [Result] Markovic G, Mikulic P. Neuro-musculoskeletal and performance adaptations to lower-extremity plyometric training. Sports Med. 2010 Oct 1;40(10):859-95. doi: 10.2165/11318370-000000000-00000. PMID 20836583
- [Result] Castro-Pinero J, Ortega FB, Artero EG, Girela-Rejon MJ, Mora J, Sjostrom M, Ruiz JR. Assessing muscular strength in youth: usefulness of standing long jump as a general index of muscular fitness. J Strength Cond Res. 2010 Jul;24(7):1810-7. doi: 10.1519/JSC.0b013e3181ddb03d. PMID 20555277
- [Result] Noyes FR, Barber SD, Mangine RE. Abnormal lower limb symmetry determined by function hop tests after anterior cruciate ligament rupture. Am J Sports Med. 1991 Sep-Oct;19(5):513-8. doi: 10.1177/036354659101900518. PMID 1962720